CLINICAL TRIAL: NCT03131401
Title: Determination of the Prevalence of LF Infection in Districts Not Included in LF Control Activities and of the Basis for Integrated Implementation of LF - Onchocerciasis Elimination Strategies in Potentially Co-endemic Areas
Brief Title: Prevalence of LF Infection in Districts Not Included in LF Control Activities
Status: Completed | Type: Observational
Sponsor: Noguchi Memorial Institute for Medical Research (Other)
Collaborators: Ghana Health Service, Neglected Tropical Diseases Program (Other)
Responsible Party: Sponsor
Other Study IDs: TDR B40376
Record Dates: First submitted 2017-02-27; First posted 2017-04-27 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Lymphatic Filariases; Onchocerciasis
MeSH Terms: conditions — Elephantiasis, Filarial; Onchocerciasis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Only parasite positive blood specimen and DNA will be retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Diagnostic Test: Diagnosis of lymphatic filariasis — Field validation of the diagnostic performance of diagnostic tests for infection with W. bancrofti.
  Other Names: Filaria Test Strip; Wb123 RDT
Diagnostic Test: Diagnosis of lymphatic Filariasis and onchocerciasis — Field validation of the diagnostic performance of diagnostic tests for infection with both W. bancrofti and O. volvulus.
  Other Names: Wb123-Ov16 RDT
Diagnostic Test: DEC Patch — Field validation of the diagnostic performance of diagnostic tests for infection with O. volvulus.
  Other Names: Diagnosis of onchocerciasis

SUMMARY:
Lymphatic filariasis is a neglected tropical disease earmarked for elimination as a public health problem by the year 2020. Since the year 2000, the Global Program for the Elimination of LF has together with endemic countries undertaken preventive chemotherapy in endemic districts to entire at risk populations. In Ghana, treatment of LF is based on the drugs Ivermectin and Albendazole. Remarkable achievements have been made towards the control and elimination of LF in Ghana. However, there remain programmatic and implementation challenges that need to be addressed in order to ensure that the gains made over the last 15 years are sustained. Among these challenges is the persistent transmission of LF in some districts despite more than 10 years of MDA.

Furthermore, LF cases have been identified in communities from eight districts, previously considered as non-endemic. The extent of endemicity in these new districts is unknown. In order to achieve the 2020 elimination targets, it is crucial to determine the distribution and infection prevalence of LF in these districts. Evaluating these districts for LF endemicity will help the implementation of appropriate strategies towards achieving the 2020 target.

This protocol describes the surveys to be undertaken in Ghana in 3 of these districts. The current standard mapping methodologies of LF have the potential to miss LF endemic villages, due to the focal nature of LF. As such, in order to enhance the chances to detect endemic communities, this survey will use a combination of the WHO EPI cluster survey and current LF mapping protocols. 15 communities will be selected in each district, with 100 survey participants per community. Survey participants will be screened for LF infection using immunological and parasitological methods. Study participants will also be tested for onchocerciasis infection using immunological and parasitological methods in districts where LF and oncho are co-endemic. The information from this survey will be combined with the data on the LF vectors and their infection status in the survey areas and relevant data available at the Ghana Health Service to:

1. determine whether LF intervention strategies are indicated in these three districts,
2. design, as indicated, appropriate intervention strategies to achieve LF elimination in these three districts by 2020
3. inform, if indicated, co-implementation of control, monitoring and evaluation for LF and onchocerciasis in the two onchocerciasis endemic districts
4. extract lessons learnt for the design and implementation of surveys in the other districts currently considered non-endemic but where LF cases have been reported.

New rapid diagnostic tests have been developed to assess infection Lf and onchocerciasis infection prevalence at the time of the decision to stop MDA and for surveillance for new infections once MDA has been stopped. These include Rapid Diagnostic Tests (RDT) for antibodies against the W. bancrofti antigen WB123 and the O. volvulus antigen Ov16. These tests still require large scale field validation. Provided additional funding becomes available, this survey will be used to obtain field validation data.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to provide informed consent (or assent with parental/guardian consent)
* Age ≥ 5 years
* Residency in the study villages since birth or for at least the previous five years

Exclusion Criteria:

* Inability to come out of bed
* Feeling sick
* Inability to provide consent

Min Age: 5 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted in districts considered non-endemic for LF based on the Ghana wide LF mapping conducted in 2000, but where LF cases have been identified. These districts fall within the Eastern and Volta Regions. At least one district has been selected in each of these regions. The selected study districts are East Akim, Hohoe and Adaklu. East Akim and Hohoe districts are also endemic for onchocerciasis.
Sampling Method: Probability Sample
Enrollment: 3736 (Actual)
Dates: Start 2018-01-21 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of lymphatic Filariasis | 3 months
  To determine the prevalence and distribution of LF infection in three districts previously considered non-endemic but reporting LF cases
Measures of protection | 3 months
  To determine what measures the population in these districts use to protect themselves from mosquito bites
Prevalence on Onchocerciasis | 3 months
  To determine the prevalence and intensity of infection with O. volvulus in two of these three districts known to be onchocerciasis endemic
Vectors of lymphatic Filariasis | 6 months
  To determine the LF vectors in three districts considered non-endemic for LF
Wuchereria bancrofti infection in vectors | 12 months
  To assess the prevalence of W. bancrofti infection in mosquitoes in these districts.

SECONDARY OUTCOMES:
Performance of diagnostic tests | 12 months
  To characterize the diagnostic performance via the standard parameters sensitivity and specificity of different diagnostic tests

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Boakye, PhD, Principal Investigator — Noguchi Memorial Institute for Medical Research
Locations (1):
- Villages in Eastern and Volta Region, Eastern and Volta Regions, Ghana

IPD SHARING:
Plan to Share IPD: No